CLINICAL TRIAL: NCT07370948
Title: Study of the Antibiotic-resistance Profile of Enterobacterales Isolated From Rectal Mucosal Buffer of PrEP Subjects
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ENTERO-PrEP
Record Dates: First submitted 2025-12-17; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- male and female subjects aged between 18 and 45 years who use PrEP: male and female subjects aged between 18 and 45 years who use PrEP and who go to the dedicated clinics of the Infectious Diseases Unit of the IRCCS - University Hospital of Bologna for normal follow-up visits Patients will be treated in accordance with their normal care process and the results of the study-specific laboratory analyses provided for by this protocol will in no way influence the diagnostic-therapeutic path of the patients.

SUMMARY:
The importance of the study lies mainly in expanding knowledge of the phenomenon of antibiotic resistance in subjects using PrEP, studying for the first time in this population the resistance phenotype in commensal Enterobacterales of the gastrointestinal tract.

The data obtained from this study could pave the way for potential surveillance and awareness programs for the critical and conscious use of antimicrobials in PrEP subjects in order to mitigate the problem of antibiotic resistance, which currently represents a real global challenge.

DETAILED DESCRIPTION:
ENTERO-PrEP is an observational, single-center, cross-sectional, tissue study. Patient enrollment will be performed at dedicated clinics for the monitoring and follow-up of PrEP subjects at the Infectious Diseases Unit of the IRCCS - University Hospital of Bologna.

In these clinics, on a quarterly basis, PrEP subjects undergo, as a normal diagnostic-assistance path, laboratory tests to exclude the presence of STIs, including the search for Chlamydia trachomatis and Neisseria gonorrhoeae in genital (urine) and extra-genital samples (pharyngeal swab and anorectal swab).

Each patient will be recruited only once during one of the normal monitoring visits scheduled for subjects using PReP.

The study aims to isolate commensal Enterobacterales strains from the gastrointestinal tract starting from the same anorectal swab sent for the detection of C. trachomatis and N. gonorrhoeae, without the need to perform any additional sampling compared to the normal care routine. For each isolated Enterobacterales strain, the sensitivity/resistance to antimicrobials (antibiogram) will subsequently be studied using broth micro-dilution. Bacterial isolation and antibiogram will be performed at the Microbiology Unit of the IRCCS - University Hospital of Bologna.

Subjects who consent to participate in the study will be asked to complete, directly during the outpatient visit, a questionnaire with information relating to personal and behavioral habits in order to identify risk factors that could favor the presence of antibiotic-resistant Enterobacterales.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 45 years
* HIV-negative subjects undergoing an anorectal swab for Chlamydia trachomatis and Neisseria gonorrhoeae using NAAT as a normal diagnostic-assistance procedure provided for subjects using PrEP

Exclusion Criteria:

* none

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: male and female subjects aged between 18 and 45 years who use PrEP and who go to the dedicated clinics of the Infectious Diseases Unit of the IRCCS - University Hospital of Bologna for normal check-ups/follow-ups Patients will be treated in accordance with their normal care process and the results of the study-specific laboratory analyses provided for by this protocol will in no way influence the diagnostic-therapeutic path of the patients.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Prevalence of antibiotic-resistant Enterobacterales strains | At enrolment
  Percentage of resistant strains out of the total strains isolated for each individual antimicrobial based on MICs obtained by a phenotypic antibiogram in broth micro-dilution, compared with criteria by EUCAST guidelines (www.eucast.org/).

SECONDARY OUTCOMES:
Prevalence of antibiotic-resistant Enterobacterales strains | At enrolment
  Percentage of resistant strains out of the total strains isolated for each individual antimicrobial based on MICs obtained by a phenotypic antibiogram in broth micro-dilution, compared with criteria by EUCAST guidelines (www.eucast.org/).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams ADN, Wood F, Gillespie D, Couzens Z, Hughes K, Hood K. The relationship between HIV pre-exposure prophylaxis, sexually transmitted infections, and antimicrobial resistance: a qualitative interview study of men who have sex with men. BMC Public Health. 2022 Nov 29;22(1):2222. doi: 10.1186/s12889-022-14645-0. PMID 36447181
- [Background] Van Dijck C, Laumen JGE, de Block T, Abdellati S, De Baetselier I, Tsoumanis A, Malhotra-Kumar S, Manoharan-Basil SS, Kenyon C, Xavier BB. The oropharynx of men using HIV pre-exposure prophylaxis is enriched with antibiotic resistance genes: A cross-sectional observational metagenomic study. J Infect. 2023 Apr;86(4):329-337. doi: 10.1016/j.jinf.2023.02.006. Epub 2023 Feb 9. PMID 36764395
- [Background] Vanbaelen T, Van Dijck C, De Baetselier I, Florence E, Reyniers T, Vuylsteke B, Jacobs BK, Kenyon C. Screening for STIs is one of the main drivers of macrolide consumption in PrEP users. Int J STD AIDS. 2021 Oct;32(12):1183-1184. doi: 10.1177/09564624211025940. Epub 2021 Jun 17. No abstract available. PMID 34139924
- [Background] Traeger MW, Schroeder SE, Wright EJ, Hellard ME, Cornelisse VJ, Doyle JS, Stoove MA. Effects of Pre-exposure Prophylaxis for the Prevention of Human Immunodeficiency Virus Infection on Sexual Risk Behavior in Men Who Have Sex With Men: A Systematic Review and Meta-analysis. Clin Infect Dis. 2018 Aug 16;67(5):676-686. doi: 10.1093/cid/ciy182. PMID 29509889
- [Background] Quaife M, MacGregor L, Ong JJ, Gafos M, Torres-Rueda S, Grant H, Terris-Prestholt F, Vickerman P. Risk compensation and STI incidence in PrEP programmes. Lancet HIV. 2020 Apr;7(4):e222-e223. doi: 10.1016/S2352-3018(19)30333-9. Epub 2019 Nov 22. No abstract available. PMID 31767536
- [Background] Perez-Galera S, Bravo-Ferrer JM, Paniagua M, Kostyanev T, de Kraker MEA, Feifel J, Sojo-Dorado J, Schotsman J, Canton R, Daikos GL, Carevic B, Dragovac G, Tan LK, Raka L, Hristea A, Viale P, Akova M, Reguera JM, Valiente de Santis L, Torre-Cisneros J, Cano A, Roilides E, Radulovic L, Kirakli C, Shaw E, Falagas ME, Pintado V, Goossens H, Bonten MJ, Gutierrez-Gutierrez B, Rodriguez-Bano J; COMBACTE-CARE-EURECA Team. Risk factors for infections caused by carbapenem-resistant Enterobacterales: an international matched case-control-control study (EURECA). EClinicalMedicine. 2023 Feb 27;57:101871. doi: 10.1016/j.eclinm.2023.101871. eCollection 2023 Mar. PMID 36895801
- [Background] Ong JJ, Baggaley RC, Wi TE, Tucker JD, Fu H, Smith MK, Rafael S, Anglade V, Falconer J, Ofori-Asenso R, Terris-Prestholt F, Hodges-Mameletzis I, Mayaud P. Global Epidemiologic Characteristics of Sexually Transmitted Infections Among Individuals Using Preexposure Prophylaxis for the Prevention of HIV Infection: A Systematic Review and Meta-analysis. JAMA Netw Open. 2019 Dec 2;2(12):e1917134. doi: 10.1001/jamanetworkopen.2019.17134. PMID 31825501
- [Background] Mogaka FO, Stewart J, Omollo V, Bukusi E. Challenges and Solutions to STI Control in the Era of HIV and STI Prophylaxis. Curr HIV/AIDS Rep. 2023 Oct;20(5):312-319. doi: 10.1007/s11904-023-00666-w. Epub 2023 Sep 26. PMID 37751130
- [Background] Miller WR, Arias CA. ESKAPE pathogens: antimicrobial resistance, epidemiology, clinical impact and therapeutics. Nat Rev Microbiol. 2024 Oct;22(10):598-616. doi: 10.1038/s41579-024-01054-w. Epub 2024 Jun 3. PMID 38831030
- [Background] McCormack S, Dunn DT, Desai M, Dolling DI, Gafos M, Gilson R, Sullivan AK, Clarke A, Reeves I, Schembri G, Mackie N, Bowman C, Lacey CJ, Apea V, Brady M, Fox J, Taylor S, Antonucci S, Khoo SH, Rooney J, Nardone A, Fisher M, McOwan A, Phillips AN, Johnson AM, Gazzard B, Gill ON. Pre-exposure prophylaxis to prevent the acquisition of HIV-1 infection (PROUD): effectiveness results from the pilot phase of a pragmatic open-label randomised trial. Lancet. 2016 Jan 2;387(10013):53-60. doi: 10.1016/S0140-6736(15)00056-2. Epub 2015 Sep 9. PMID 26364263
- [Background] Li H, Liu B, Li M, Shen M. Livestock and poultry breeding farms as a fixed and underestimated source of antibiotic resistance genes. Environ Sci Pollut Res Int. 2024 Aug;31(37):49916-49931. doi: 10.1007/s11356-024-34413-4. Epub 2024 Jul 25. PMID 39052112
- [Background] Laumen JGE, Van Dijck C, Abdellati S, De Baetselier I, Serrano G, Manoharan-Basil SS, Bottieau E, Martiny D, Kenyon C. Antimicrobial susceptibility of commensal Neisseria in a general population and men who have sex with men in Belgium. Sci Rep. 2022 Jan 7;12(1):9. doi: 10.1038/s41598-021-03995-1. PMID 34997050
- [Background] Kenyon C. Dual Azithromycin/Ceftriaxone Therapy for Gonorrhea in PrEP Cohorts Results in Levels of Macrolide Consumption That Exceed Resistance Thresholds by up to 7-Fold. J Infect Dis. 2021 Nov 16;224(9):1623-1624. doi: 10.1093/infdis/jiab178. No abstract available. PMID 33822092
- [Background] Huang KD, Amend L, Galvez EJC, Lesker TR, de Oliveira R, Bielecka A, Blanco-Miguez A, Valles-Colomer M, Ruf I, Pasolli E, Buer J, Segata N, Esser S, Strowig T, Kehrmann J. Establishment of a non-Westernized gut microbiota in men who have sex with men is associated with sexual practices. Cell Rep Med. 2024 Mar 19;5(3):101426. doi: 10.1016/j.xcrm.2024.101426. Epub 2024 Feb 15. PMID 38366600
- [Background] Cai S, Wang Z, Han X, Hu H, Quan J, Jiang Y, Du X, Zhou Z, Yu Y. The correlation between intestinal colonization and infection of carbapenem-resistant Klebsiella pneumoniae: A systematic review. J Glob Antimicrob Resist. 2024 Sep;38:187-193. doi: 10.1016/j.jgar.2024.04.013. Epub 2024 May 21. PMID 38777180